CLINICAL TRIAL: NCT03095040
Title: The Efficacy and Safety of CM082 Combined With Everolimus in Chinese Patients With Metastatic Renal Cell Carcinoma: a Randomized, Double-blind, Double Dummy, Multicenter Study
Brief Title: CM082 Combined With Everolimus in Chinese Patients With Metastatic Renal Cell Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CM082-CA-Ⅱ-201
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Renal Cell Cancer Metastatic
MeSH Terms: interventions — Everolimus; vorolanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CM082 combined with everolimus (Experimental)
  Interventions: Drug: CM082 combined with everolimus
- CM082 (Experimental)
  Interventions: Drug: CM082
- Everolimus (Active Comparator)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: CM082 combined with everolimus — CM082 tablets (200 mg, 2 tablets) taken orally once a day on 28-day cycles, everolimus tablets (10 mg, 2 tablets) taken orally once a day on 28-day cycles
  Other Names: X-82; Affinitor
  Arms: CM082 combined with everolimus
Drug: CM082 — CM082 tablets (200 mg, 2 tablets) taken orally once a day on 28-day cycles, dummy tablets for everolimus (2 tablets) taken orally once a day on 28-day cycles
  Other Names: X-82
  Arms: CM082
Drug: Everolimus — Everolimus tablets (10 mg, 2 tablets) taken orally once a day on 28-day cycles, dummy tablets for CM082 (2 tablets) taken orally once a day on 28-day cycles
  Other Names: Affinitor
  Arms: Everolimus

SUMMARY:
This randomized, double blind, phase 2/3 study is aimed to evaluate the efficacy and safety of CM082 in combination with everolimus in Chinese patients with advanced renal cell carcinoma. The primary endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of clear cell renal cell carcinoma
* Progressed on at least one standard therapy with VEGFR TKI
* Measurable disease per Recist v1.1
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1
* Life expectancy of at least 12 weeks
* Adequate organ functions, and meet the following requirements:

Bone marrow: ANC ≥1.5*109/L (1500/mm3), platelet ≥100*109/L, and hemoglobin ≥9 g/dL Liver: Total bilirubin ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5x the upper limit of normal (ULN) if no liver involvement or ≤5x the upper limit of normal with liver involvement Kidney: Creatinine ≤ 1.25 x ULN, urine protein <1+ Heart: LVEF ≥ 50%

* Willingness and ability to comply with trial and follow-up procedures
* Ability to understand the nature of this trial and give written informed consent

Exclusion Criteria:

* Currently receiving anti-cancer treatment; currently or previously have received 2 or more systemic anti-cancer treatment
* Other tumors in addition to renal cell carcinoma
* Females who are pregnant or breastfeeding
* Known hypersensitivities to CM082 or everolimus
* Those with concurrent condition(e.g. psychological, neuronal, cardiovascular, respiratory conditions or infections) that in the investigator's opinion would jeopardize compliance with the protocol
* Patients with known central nervous system (CNS) metastases
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of CM082 or everolimus
* Any active infection
* Drug or alcohol abuser

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2016-12-16 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  The internal between the date of randomization and the date of disease progression, unaccepted toxicity, or death

SECONDARY OUTCOMES:
Overall survival | 36 months
  The internal between the date of randomization and the date of death
Objective response rate | 8 weeks
  The percentage of patients with tumor response in overall population

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheng X, Ye D, Zhou A, Yao X, Luo H, He Z, Wang Z, Zhao Y, Ji Z, Zou Q, He C, Guo J, Tu X, Liu Z, Shi B, Liu B, Chen P, Wei Q, Hu Z, Zhang Y, Jiang K, Zhou F, Wu D, Fu C, Li X, Wu B, Wang L, Qin S, Li G, Liu Y, Guo H, Chen K, Zhang D, Wang G, Ding L, Wang Y, Yuan X, Guo J. Efficacy and safety of vorolanib plus everolimus in metastatic renal cell carcinoma: A three-arm, randomised, double-blind, multicentre phase III study (CONCEPT). Eur J Cancer. 2023 Jan;178:205-215. doi: 10.1016/j.ejca.2022.10.025. Epub 2022 Nov 1. PMID 36459768
- [Derived] Sheng X, Yan X, Chi Z, Cui C, Si L, Tang B, Li S, Mao L, Lian B, Wang X, Bai X, Zhou L, Kong Y, Dai J, Ding L, Mao L, Guo J. Phase 1 trial of vorolanib (CM082) in combination with everolimus in patients with advanced clear-cell renal cell carcinoma. EBioMedicine. 2020 May;55:102755. doi: 10.1016/j.ebiom.2020.102755. Epub 2020 Apr 23. PMID 32335374